CLINICAL TRIAL: NCT05793294
Title: Nutritional Status, Health and Gut Microbiome Development in Children; a Prospective Cohort Study From Pakistan
Brief Title: Child Health, Nutrition and Microbiome Development
Acronym: CHAMP
Status: Active, not recruiting | Type: Observational
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: University of Reading (Other); Abdul Wali Khan University Mardan (Other); University of Bern (Other); National Institute of Health, Pakistan (Unknown)
Responsible Party: Sponsor
Other Study IDs: Gut microbiome development; NHCG-22/R2-74 (Other Grant/Funding Number: National Institute of Health, Pakistan)
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Malnutrition; Stunting; Wasting; Underweight; Overweight and Obesity
Keywords: Nutritional status; Gut microbiome; Health; Anthropometry; Malnutrition; Stunting; Wasting; Underweight; Overweight; Growth
MeSH Terms: conditions — Malnutrition; Growth Disorders; Cachexia; Thinness; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Serum, plasma, and stool samples will be stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Birth cohort: All infants age 0 - 28 days will be recruited and followed until 24 months of age

SUMMARY:
Childhood malnutrition is a global public health issue with devastating consequences on the health, well-being, and psychosocial development of children. Emerging evidence suggests that malnourished children have immature gut microbiota compared to age-matched healthy controls and it does not repair even after nutritional interventions. The present study aims to characterize how the gut microbiome develops during the first two years of life in children residing in malnutrition endemic areas of Khyber Pakhtunkhwa, the region with the highest prevalence of childhood malnutrition in Pakistan and the region.

DETAILED DESCRIPTION:
Malnutrition in children remains a global public health challenge. The consequences are often severe and deadly, particularly in low- and middle-income countries where malnutrition contributes to ~half of deaths in children under five years of age. Pakistan is among those nations with the highest burden of stunting (40.2%), wasting (17.7%), and micronutrient deficiency in children under five years of age. Recently, scientists discovered that the trillions of microbes (gut microbiome) that live in the human gut affect the nutritional status and overall health of children during the initial years of life. In this context, research studies from developing countries, where malnutrition is common, have reported an impaired or immature gut microbiome in malnourished (stunted, wasted, and underweight) children compared to matched healthy controls and it does not repair even after nutritional intervention. Therefore, a nutritional intervention strategy that does not take into account the gut microbiome microbiota will fail to ameliorate the long-term consequences of malnutrition.

In this prospective cohort study from Pakistan, healthy infants (n=70) aged 0 - 28 days will be recruited from rural and remote areas of District Swat and followed at 3, 6, 12, 18 and 24 months. Ante-natal and postnatal history, Dietary intake data, dietary diversity, Infant and young child feeding (IYCF practices), and Health outcomes data will be collected at baseline and followup. The investigators will also collect dry blood spot, stool and oral swab samples and conduct anthropometric assessments of both mother and the baby at each time point. Advanced, next-generation sequencing technology will be used to explore gut microbiome diversity and functional potential.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 0 - 28 days
* Born to parents residing in rural and remote areas of District Swat
* Living in separate households
* Parents/caregivers have no plans to move out of the stud site for at least one year after enrollment in the study.

Exclusion Criteria:

* Child born to underage (<18 years old) mother.
* Infants born with severe acute or chronic medication conditions that require hospitalization or prolonged use of medication or both or the infant is diagnosed with enteropathies.
* Whose parents refused to provide informed consent to participate in the study.
* Weight of the child is <1500 gm.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The eligible participants (neonates) will be identified by searching the health and immunization record of the recently born children in the study area. The record will be obtained from the health facilities serving the study area. Eligible participants will be recruited with the help of trained Lady Health Workers.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome profile | 2 years
  Next generation sequencing to asses changes in gut microbiome diversity and functional potential at 0, 3, 6, 9, 12, 18 and 24 months of age. These data will then be categorised on the basis of nutritional status (Healthy, Stunting, Wasting), dietary patterns and health status.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shahzad, PhD, Principal Investigator — Khyber Medical University; Zia Ul Haq, PhD, Study Director — Khyber Medical University
Locations (2):
- Pakistan (2):
  - Khyber Medical University, Peshawar, Khyber Pakhtunkhwa
  - Tehsil Matta, Swāt, Khyber Pakhtunkhwa

IPD SHARING:
Plan to Share IPD: No